CLINICAL TRIAL: NCT02705508
Title: Phase 2 Trial of PEG-ASP Combined With Etoposide and Gemcitabine (PEG) as First-line Chemotherapy to Treat NK/T-cell Lymphoma
Brief Title: PEG-ASP, Etoposide and Gemcitabine for Natural Killer/T Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, Hua Wang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-SYSUCC-2016
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Treatment Refusal
Keywords: extranodal natural killer/T-cell lymphoma; nasal type; chemotherapy; radiotherapy
MeSH Terms: conditions — Treatment Refusal | interventions — Gemcitabine; Etoposide; etoposide phosphate; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG group (Experimental): Treatment PEG dosages were as follows: days 1 and 8,30min intravenous infusion of 1000mg/m2 gemcitabine;day1,4h intravenous infusion of 100mg/m2 etoposide,day1-3,deep intramuscular injection of 2500U/m2 Pegaspargase at three different sites.The regimen was repeated every 3 weeks.Stage IE/IIE patients underwent four cycles induction chemotherapy, followed by involved-field radiotherapy after got CR, PR or SD. Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved-field radiation (IFRT) dose was 50-56 Gy.Stage IIIE/IVE patients were given for a maximum of six cycles.
  Interventions: Drug: Gemcitabine; Drug: etoposide; Drug: Pegaspargase; Radiation: involved-field radiotherapy

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2, ivd on day 1 and 8 of each 21 day cycle.
  Other Names: Gemzar
Drug: etoposide — 100mg/m2，4h-intravenous infusion on day1-3 of each 21 day cycle.
  Other Names: Etoposide phosphate
Drug: Pegaspargase — 2500U/m2 im on day 1 of each 21 day cycle.
  Other Names: Oncaspar
Radiation: involved-field radiotherapy — Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved- field radiation (IFRT) dose was 50-56 Gy.
  Other Names: IFRT

SUMMARY:
Extranodal natural killer/T-cell lymphoma (ENKTL) is an aggressive form of non-Hodgkin's lymphoma and shows extremely poor survival. This prospective pilot study to evaluate the efficacy and safety of pegylated aspargase(PEG-ASP)combined with etoposide and gemcitabine (PEG) treatment in this population.

DETAILED DESCRIPTION:
Treatment PEG dosages were as follows: days 1 and 8,30min intravenous infusion of 1000mg/m2 gemcitabine;day1,4h intravenous infusion of 100mg/m2 etoposide,day1-3,deep intramuscular injection of 2500unit/m2 PEG-ASP at three different sites.The regimen was repeated every 3 weeks.Stage IE/IIE patients underwent four cycles induction chemotherapy, followed by involved-field radiotherapy after got complete remission ,partial regression or stable disease.Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved-field radiation (IFRT) dose was 50-56 Gy.Stage IIIE/IVE patients were given for a maximum of six cycles.Refractory/relapsed patients underwent at least two cycles treatments unless there was disease progression or unacceptable side effects, or withdrawal of patient consent. Autologous haematopoietic stem cell transplantation (AHSCT) was recommended after achieving CR for advanced stage and refractory/relapsed patients

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed, previously untreated or refractory/relapsed ENKTL as defined by the World Health Organization classification;
2. age≥18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. at least one measurable lesion;
5. adequate haematologic function (haemoglobin > 9.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l),
6. adequate hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal),
7. adequate renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min);
8. normal coagulation function and electrocardiogram results.
9. Prior chemotherapy and radiotherapy should have been completed >4 weeks 10.earlier,willingness to provide written informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)

SECONDARY OUTCOMES:
overall survival | up to end of follow-up-phase (approximately 3 years)
complete remission rate | every 3 weeks,up to completion of chemotherapy(approximately 3months)

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | up to end of follow-up-phase (approximately 3 years)
  including hematological safety and non-hematological safety

CONTACTS AND LOCATIONS:
Overall Officials: hua wang, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Please Select, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Feng D, Yan Z, Fu B, Bai S, Zhu L, Gale RP, Xia Z, Liang Y, Wang H. Phase II study of pegaspargase, etoposide, gemcitabine (PEG) followed by involved-field radiation therapy in early-stage extranodal natural killer/T-cell lymphoma. Hematology. 2024 Dec;29(1):2402102. doi: 10.1080/16078454.2024.2402102. Epub 2024 Sep 13. PMID 39268981